CLINICAL TRIAL: NCT03534154
Title: Developing and Validating Blood and Imaging BIOmarkers of AXonal Injury Following Traumatic Brain Injury
Acronym: BIO-AX-TBI
Status: Completed | Type: Observational
Sponsor: Imperial College London (Other)
Collaborators: Centre Hospitalier Universitaire Vaudois (Other); University College, London (Other); Istituto Di Ricerche Farmacologiche Mario Negri (Other); Fondazione IRCCS Ca' Granda, Ospedale Maggiore Policlinico (Other)
Responsible Party: Sponsor
Other Study IDs: 230221; MR/R004528/1 (Other Grant/Funding Number: ERA-NET)
Record Dates: First submitted 2018-04-27; First posted 2018-05-23 (Actual); Last update posted 2022-03-31 (Actual); Status verified 2022-03

CONDITIONS: Traumatic Brain Injury
MeSH Terms: conditions — Brain Injuries, Traumatic | interventions — Blood Specimen Collection; Magnetic Resonance Imaging

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Blood and cerebral microdialysis samples collected during longitudinal study, where appropriate (as per protocol).
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- TBI - MRI / bloods / cognitive / clinical outcomes: Work package 1. In a large multi-centre cohort of adult moderate/severe TBI patients we aim to identify the most informative plasma biomarker(s) of the severity of axonal injury. We will characterise their time course, focusing on neurofilament light (NFL) and tau, and relate these to magnetic resonance imaging (MRI) measures of axonal injury. Using logistic regression we will then test whether these measures contribute to the prediction of clinical outcome at twelve months
  Interventions: Diagnostic Test: MRI; Diagnostic Test: Blood Sampling; Diagnostic Test: Neuropsychological tests
- TBI - Advanced MRI / bloods / cognitive / clinical outcomes: Work package 2. In a subgroup of the patients recruited to WP1 we will use advanced MRI and longitudinal assessments to provide a more detailed description of the relationship between the plasma biomarkers and outcome after TBI. We will test whether advanced diffusion and myelin integrity measures correlate with plasma biomarkers and whether early plasma biomarker levels predict neurodegeneration measured by progressive atrophy after TBI.
  Interventions: Diagnostic Test: MRI; Diagnostic Test: Blood Sampling; Diagnostic Test: Neuropsychological tests; Diagnostic Test: MRI (advanced)
- TBI - microdialysis / adv. MRI / cognitive / clinical: Work package 3. In a second subgroup of patients recruited to WP1 we will combine microdialysis, neuroimaging and plasma sampling of axonal proteins to provide a deeper understanding of the mechanisms of axonal injury progression and use this approach to investigate the axonal origin of the plasma biomarkers.
  Interventions: Diagnostic Test: MRI; Diagnostic Test: Blood Sampling; Diagnostic Test: Microdialysis; Diagnostic Test: Neuropsychological tests; Diagnostic Test: MRI (advanced)
- Healthy volunteer: Single assessment using MRI, bloods and cognitive testing.
  Interventions: Diagnostic Test: MRI; Diagnostic Test: Blood Sampling; Diagnostic Test: Neuropsychological tests

INTERVENTIONS:
Diagnostic Test: MRI — Magnetic Resonance Imaging
Diagnostic Test: Blood Sampling — Sampling of serum
Diagnostic Test: Microdialysis — Monitoring of cerebral fluid protein levels
  Groups: TBI - microdialysis / adv. MRI / cognitive / clinical
Diagnostic Test: Neuropsychological tests — Battery of tests to assess cognitive function, patient outcomes
Diagnostic Test: MRI (advanced) — Advanced MRI
  Groups: TBI - Advanced MRI / bloods / cognitive / clinical outcomes; TBI - microdialysis / adv. MRI / cognitive / clinical

SUMMARY:
Observational longitudinal study assessing outcomes following moderate-severe traumatic brain injury (TBI).

DETAILED DESCRIPTION:
Traumatic brain injury (TBI) occurs when the brain is physically damaged, for example after a car crash. It is common and survivors often have major on-going problems. It is very difficult to predict how patients will do after TBI. One reason for this is that clinicians and researchers are unable to measure all the effects of TBI. An important factor is that the connections between nerve cells are damaged by the impact on the brain of an injury (axonal injury). This damage has been difficult to measure in the past, but new ways to scan the brain and more sensitive ways of picking up the effects of this injury in the blood could change this. In other parts of medicine tests of this type have had a dramatic effect on how clinicians treat patients. For example, the products of heart muscle damage that have leaked into the blood can be used identify a heart attack and guide treatment. Clinicians need similar tests to be available in TBI. This should be possible as the products of axonal injury also leak into the blood and researchers have a sensitive way to pick this up. An accurate test for axonal injury would guide treatment choices and allow clinicians to predict how patients will recover. The investigators have brought together an international team who have been working on different aspects of this problem for many years. Together the investigators will conduct a large study to identify the best measures of axonal injury. The investigators will carefully test whether these measures help predict outcomes and will study where the blood markers come from using a safe method to measure the effects of axonal injury directly from the brain. The work links into some large projects that have already started and will use a standard way to assess patients after their injury. This is important because it will allow researchers to share results across studies. The investigators hope the work will allow us to identify a blood marker for TBI that could be widely used to quickly identify the presence of axonal injury. The investigators will also show what brain imaging measure is best at picking up axonal injury and how best to combine the measures to best predict how patients recover. This will allow doctors to diagnose problems after TBI more accurately, choose the right treatments and give patients and their families accurate advice about what will happen after discharge from hospital.

ELIGIBILITY:
Inclusion Criteria:

* A diagnosis of moderate/severe traumatic brain injury (TBI) as classified using the Mayo classification system;
* Healthy controls will be age-matched to our TBI patients and will not have a history of significant neurological or psychiatric conditions.

Exclusion Criteria:

* Unwillingness or inability to follow the procedures required
* Bilateral fixed dilated pupils
* For MRI, contra-indication to MRI scanning, assessed by a standard pre-MRI questionnaire (e.g. presence of ferromagnetic implants in the body, claustrophobia, pregnancy) if considered for the imaging strand of the study.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: 250 traumatic brain injury patients from ITU / major trauma ward.
Sampling Method: Non-Probability Sample
Enrollment: 313 (Actual)
Dates: Start 2017-11-30 (Actual); Primary Completion 2021-04-30 (Actual); Study Completion 2021-12-30 (Actual)

PRIMARY OUTCOMES:
Change in diffusion tensor imaging measures over time | 10 days - 6 weeks, 6 months and 12 months
  Fractional anisotropy (FA)
Brain atrophy rates | 10 days - 6 weeks, 6 months and 12 months
  Brain tissue volume changes over time.
Change in levels of fluid biomarkers in blood | 0-5 days, 5-10 days, 10 days - 6 weeks, 6 months and 12 months
  Neurofilament light and Tau protein
Change in levels of fluid biomarkers in cerebral fluid | 48 hours to 7 days
  Neurofilament light and Tau protein

CONTACTS AND LOCATIONS:
Overall Officials: David Sharp, Principal Investigator — Imperial College London
Locations (5):
- Italy (2):
  - Fondazione IRCCS, Ca' Granda Ospedale Maggiore Policlinico, Milan
  - IRCCS - Istituto di Ricerche Farmacologiche "Mario Negri", Milan
- University Medical Centre, Ljubljana, Slovenia
- Centre Hospitalier Universitaire Vaudois, Lausanne, Switzerland
- Imperial College London, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Graham NSN, Zimmerman KA, Bertolini G, Magnoni S, Oddo M, Zetterberg H, Moro F, Novelli D, Heslegrave A, Chieregato A, Fainardi E, Fleming JM, Garbero E, Abed-Maillard S, Gradisek P, Bernini A, Sharp DJ. Multicentre longitudinal study of fluid and neuroimaging BIOmarkers of AXonal injury after traumatic brain injury: the BIO-AX-TBI study protocol. BMJ Open. 2020 Nov 10;10(11):e042093. doi: 10.1136/bmjopen-2020-042093. PMID 33172948